CLINICAL TRIAL: NCT06529952
Title: Comparative Study Between Hysteroscopic Management of Cesarean Scar Defect and Hormonal Treatment. A Randomized Controlled Trial
Brief Title: Comparative Study Between Hormonal and Hysteroscopic Management of Cesarean Scar Defect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0107228
Record Dates: First submitted 2024-07-27; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2022-06

CONDITIONS: Cesarean Scar Defect
Keywords: cesarean scar defect; hormonal treatment; hysterscopic treatment; endocoagulation; hysteroscopic resection

STUDY DESIGN:
Intervention Model Description: the study include three groups group 1: hysterostopic resection of the upper and lower edges of the CSD then endocoagulation group2: hysteroscopic endocoagulation group3: hormonal treatment by 3rd generation contraceptive pills for 6 months
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hysteroscopic resection (Experimental): 26 patients subjected to hysteroscopic surgery in the form of resection of lower edge, resection of upper edge and endocoagulation to fulgurate the visible dilated blood vessels or endometrial-like glands inside the base of the niche by using a roller ball resectoscope with monopolar electrical current and glycine as distension media.
  Interventions: Procedure: hysteroscopic surgery by resection and endocoagulation
- hysteroscopic endocoagulation (Experimental): include 26 patients subjected to hysteroscopic endocoagulation to the base of the niche by roller ball using monopolar electrical current and glycine as distension media.
  Interventions: Procedure: hysteroscopic surgery by endocoagulation only
- hormonal treatment (Experimental): 26 patients received hormonal treatment in the form of 3rd generation combined oral contraceptive pills in a cyclic manner for 6 months.
  Interventions: Drug: hormonal treatment

INTERVENTIONS:
Procedure: hysteroscopic surgery by resection and endocoagulation — resection of lower edge, resection of upper edge and endocoagulation
  Arms: Hysteroscopic resection
Procedure: hysteroscopic surgery by endocoagulation only — hysteroscopic endocoagulation to the base of the niche by roller ball
  Arms: hysteroscopic endocoagulation
Drug: hormonal treatment — using 3rd generation contraceptive pills
  Arms: hormonal treatment

SUMMARY:
Up to 70% of women who have had a previous caesarean section experience uterine niche, with 30% having symptoms. Prevalence rates vary between 24-70% using transvaginal ultrasonography and 56-84% using gel/saline instillation sonohysterography. Classification involves the ratio of myometrial thickness at the scar to adjacent myometrium, with severe deficiency defined by a ratio of ≤50%. Dehiscence is defined as at least 80% myometrial thinning.

The aim of this work was to compare between the effectiveness of two different techniques of hysteroscopic ablation of cesarean scar defect and hormonal treatment to improve abnormal uterine bleeding and pelvic pain localized in the suprapubic area associated with isthmocele.

DETAILED DESCRIPTION:
The study include 78 women diagnosed with abnormal uterine bleeding (AUB). All cases were subjected for complete history taking, complete general and gynaecological examination, vaginal ultrasonography (TVUS) to confirm niche and exclude other pathologies. The women were randomly divided by1:1:1 ratio into three equal groups using double blind method with closed envelopes

Group A: include 26 patients subjected to hysteroscopic surgery in the form of resection of lower edge, resection of upper edge and endocoagulation to fulgurate the visible dilated blood vessels or endometrial-like glands inside the base of the niche by using a roller ball resectoscope with monopolar electrical current and glycine as distension media.

Group B: include 26 patients subjected to hysteroscopic endocoagulation to the base of the niche by roller ball using monopolar electrical current and glycine as distension media.

Group C: include 26 patients received hormonal treatment in the form of 3rd generation combined oral contraceptive pills in a cyclic manner for 6 months.

Follow up was done after 1, 3, 6 months, by TVUS to exclude presence of symptoms of abnormal uterine bleeding (AUB) and to assess different outcome measures including presence or absence of intermenstrual spotting, presence or absence of postcoital bleeding, presence or absence of Pelvic tenderness or dyspareunia

ELIGIBILITY:
Inclusion Criteria:

* women with age ranging from 25 to 42 years,
* previous cesarean section,
* presence of a cesarean scar defect on ultrasound with a residual myo3metrium of > 1.5 mm.

Exclusion Criteria:

* any contraindications of hysteroscopy as an active pelvic infection, active genital herpes,
* Contraindications to hormonal treatment as medical conditions like breast cancer, history of deep venous thrombosis, Previous arterial thrombosis, pulmonary embolism, active liver disease, use of rifampicin, familial hyperlipidemia, pregnancy,
* patient refusal
* Any Other causes of abnormal uterine bleeding as polyp, adenomyosis. leiomyoma, malignancy, coagulopathy. and ovulatory disorders.

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
presence or absence of intermenstrual spotting, | 6 months
  improvement of intermenstrual spotting in group a and B from 1 st month , and improvment in all groups after 6 months
presence or absence of postcoital bleeding | 6 months
  improvement of postcoital bleeding in all groups after 6 months
presence or absence of pelvic tenderness or dyspareunia | 6 months
  improvement of postcoital bleeding in all groups after 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - El shatby hospital Alexandria university, Alexandria
  - Tamer, Alexandria

IPD SHARING:
Plan to Share IPD: No